CLINICAL TRIAL: NCT02981732
Title: CLCF1 Gene Associated With Postmenopausal Osteoporosis of Kidney Yin Deficiency Syndrome Regulating the Bone Osteoimmunology Mechanism by the OPG/RANKL/RANK Signal System
Brief Title: CLCF1 Gene Associated With Postmenopausal Osteoporosis of Kidney Yin Deficiency Syndrome
Acronym: PMOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: xuhuijuan (Other)
Responsible Party: Sponsor-Investigator, xuhuijuan, Fujian Academy of Traditional Chinese Medicine, Fujian Academy of Traditional Chinese Medicine
Organization: Fujian Academy of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81674007
Record Dates: First submitted 2016-11-23; First posted 2016-12-05 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis; kidney yin deficiency syndrome; liuwei dihuang pill
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Shen (Kidney) yin deficiency (Experimental): Shen (Kidney) yin deficiency
  Interventions: Other: Liuwei Dihuang Pill
- the control group (No Intervention): the control group,there is no intervention

INTERVENTIONS:
Other: Liuwei Dihuang Pill
  Arms: Shen (Kidney) yin deficiency

SUMMARY:
For nearly 112 million patients with osteoporosis in China, it is of great significance for preventing and treating by clearly understanding the molecular mechanism of kidney deficiency. Thus, the research group has demonstrated in the earlier research that CLCF1 is an associated gene that can regulate JAK2/STAT3 signal pathway and impact bone metabolism for kidney yin deficiency of postmenopausal osteoporosis (PMOP). To make clear understanding of the direct-acting mechanism of CLCF1 for bone metabolism, this study intends to: ①observe impacts of low expression of CLCF1 upon immunities in mice and OPG/RANKL/RANK signal system using the technology of adenovirus associated virus. ②explore impacts of over-expression and silencing of CLCF1 on B lymphocytes by culcuturing the cells together with osteoblasts. ③ analyze the impacts of treating kidney yin deficiency of PMOP by Liuwei Dihuang pill upon immunities and OPG/RANKL/RANK system, and discuss the mechanism of regulating bone metabolism by CLCF1 by OPG/RANKL/RANK system via the bridge between immune system and bone metabolism, so as to demonstrate if the hypothesis of this study that "the molecular osteoimmunological mechanism of kidney yin deficiency of postmenopausal osteoporosis (PMOP) is possibly closely related to the impacts of CLCF1 regulation of OPG/RANKL/RANK signal system on bone metabolism" is right or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they were female Han Chinese patients who had undergone natural menopause at least 2 years prior and

  * met the diagnostic criteria for osteoporosis according to the "clinical practice guidelines of traditional medicine for primary osteoporosis"
  * met the CM diagnostic criteria according to "Syndrome Differentiation in Modern Research of Traditional Chinese Medicine"
  * provided informed consent, which was approved by the Fujian Academy of Traditional Chinese Medicine Clinical Research Ethics Committee

Exclusion Criteria:

* patients who did not meet the diagnostic criteria for osteoporosis or CM standards
* patients with rheumatoid arthritis, diabetes, secondary osteoporosis due to hyperthyroidism, and severe cardiovascular or cerebrovascular diseases
* patients with abnormal liver and/or Shen function test results
* patients with osteoporosis who had received treatment with CM within the last month, hormone replacement therapy and calcitonin within the past three months, or bisphosphonates for 15 consecutive days within the past 6 months.

Ages: 46 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
osteoporosis treatment within six months of study enrollment | Liuwei Dihuang Pills therapy(up to six months)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Academy of Trational Chiness Medicine, Fuzhou, Fujian, China